CLINICAL TRIAL: NCT06407362
Title: Evaluation of the Effects of Volume-Controlled and Pressure-Controlled Ventilation on Cerebral Oxygen Saturation, Perfusion Index, and Pleth Variability Index in Septoplasty Surgical Cases: an Observational Prospective Study
Brief Title: Effects of Volume and Pressure-Controlled Ventilation on Cerebral SpO2, PI, and PVI Index in Septoplasty
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, ahmet kaya, assistant professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: MAIEAH630001
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ventilation Mode; Pleth Variability Index; Perfusion Index; Regional Cerebral Oxygen Saturation
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had undergone septoplasty
  Interventions: Diagnostic Test: Cerebral Oxygen Saturation

INTERVENTIONS:
Diagnostic Test: Cerebral Oxygen Saturation — We have designed this study to evaluate the accuracy of PVI, PI and rSO2 in both ventilation modes in patients undergoing septorhinoplasty operation under general anaesthesia
  Other Names: Pleth Variability Index; Perfusion Index

SUMMARY:
Objective: This study was designed to evaluate the accuracy of Pleth Variability Index (PVI), Perfusion Index (PI) and Regional Oxygen Saturation (rSO2) in both ventilation modes in patients undergoing septorhinoplasty operation under general anaesthesia. Materials and Methods: After anaesthesia induction, ventilation was provided with volume control for 20 minutes. Heart Rate (HR), PI, PVI, Oxygen Saturation (SpO2), Non-Invasive Blood Pressure (NIBP) and rSO2 values were recorded every 5 minutes. At the 20th minute of the surgical procedure, the ventilation mode was set as the pressure-controlled mode. After switching to pressure-controlled mode, HR, PI, PVI, SpO2, NIBP and rSO2 values were recorded every 5 minutes for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists (ASA) score I-III between the ages of 18-80 were included

Exclusion Criteria:

* Those patients with any Liver and/or Kidney Failure
* obese patients (Body Mass Index (BMI) 30 and above)
* trauma patients
* cancer patients
* ASA IV patients
* those patients with emergency surgery
* cardiac arrhythmia
* implanted pacemakers
* those with a history of chronic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with American Society of Anesthesiologists (ASA) score I-III between the ages of 18-80 were undergoing septoplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Pleth Variability Index (PVI) in patients under different ventilation modes | while the surgery procedure
  The objective of this study was to demonstrate the percentage difference in the Pleth Variability Index (PVI) between the two ventilation modes in patients undergoing septorhinoplasty.
Perfusion Index (PI) in patients under different ventilation modes | while the surgery procedure
  The objective of this study was to demonstrate the percentage difference in the Perfusion Index (PI) between the two ventilation modes in patients undergoing septorhinoplasty.
Regional Cerebral Oxygen Saturation (rSO2) in patients under different ventilation modes | while the surgery procedure
  The objective of this study was to demonstrate the percentage difference in the Regional Cerebral Oxygen Saturation (rSO2) between the two ventilation modes in patients undergoing septorhinoplasty.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Turkey Sanliurfa Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided